CLINICAL TRIAL: NCT05095532
Title: Autologous Mesenchymal Stromal Cells and Islet Co-transplantation to Enhance Islet Survival and Function in Chronic Pancreatitis Patients Undergo Total Pancreatectomy and Islet Autotransplantation
Brief Title: Autologous Mesenchymal Stromal Cells and Islet Co-transplantation in TP-IAT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hongjun Wang, Professor, Scientific Director, Center for Cellular Therapy, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00099487; R01DK126454 (NIH)
Record Dates: First submitted 2021-10-11; First posted 2021-10-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pancreatitis; Mesenchymal Stem Cells
Keywords: Total Pancreatectomy; TP-IAT
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Intervention Model Description: This will be a randomized, controlled clinical trial in which CP patients scheduled for TP-IAT who meet the study criteria and consented will be randomized into three groups. One group will receive islet transplantation alone (n=14). The other two groups will receive islets plus BM-MSCs at two different doses (20x10^6/patient, or 50x10^6/patient, n=14 in each group).
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BM-MSCs at 20x10^6 (Experimental): One time infusion of islets plus BM-MSCs at 20x10^6/patient, n=14
  Interventions: Biological: Bone marrow-derived mesenchymal stem cells
- BM-MSCs at 50x10^6 (Experimental): One time infusion of islets plus BM-MSCs at 50x10^6/patient, n=14
  Interventions: Biological: Bone marrow-derived mesenchymal stem cells
- Placebo (Placebo Comparator): One time infusion of islets only.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Bone marrow-derived mesenchymal stem cells — MSC transplantation
  Arms: BM-MSCs at 20x10^6; BM-MSCs at 50x10^6
Other: Placebo — Standard of Care
  Arms: Placebo

SUMMARY:
This is a clinical trial for chronic pancreatitis (CP) patients undergoing total pancreatectomy with islet autotransplantation (TP-IAT). Participants will be randomized to either bone marrow-derived mesenchymal stem cells (MSCs) or control with the standard of care. Participants will be followed for one-year post-transplant.

DETAILED DESCRIPTION:
This will be a randomized, controlled clinical trial for CP patients scheduled to undergo a TP-IAT surgery. Those who are consented will be randomized into one of three groups. One group will receive islet transplantation alone, a placebo. The other two groups will receive islets plus autologous bone marrow-MSCs at two different doses (20x10^6/patient, or 50x10^6/patient). The TP-IAT procedure will remain as routinely performed. Patients will be followed for12 months post-transplantation, having 3 follow-up visits scheduled on days 90, 180, and 365 after the transplant. The primary endpoint will be a change in islet function from baseline to 12 months post-transplantation as measured by the C-peptide area under the curve following a mixed meal tolerance test. Potential effects of MSCs on glycemic control, pain relief, quality of life, and adverse events will be evaluated at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP and scheduled for TP-IAT;
* ≥18 years old;
* Diabetes with HbA1c <12%.

Exclusion Criteria:

* Patients who are under immunosuppression;
* Pregnant and breastfeeding women.
* Patients who have liver damage based on ALT, AST, and total bilirubin levels (>3 times normal levels);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Islet Cell Function | 1 year
  The primary endpoint will be change in islet function between baseline and 12 months as measured by area under the curve of C-peptide levels during a mixed meal tolerance test (MMTT) adjusted by islet equivalent number (IEQ) transplanted.

SECONDARY OUTCOMES:
Change in HbA1C levels from baseline to 12 months. | 1 year
  Change in HbA1C levels from baseline to 12 months
Proportion of insulin-independent patients following IAT | 1 year
  Proportion of insulin-independent patients following IAT
Average daily insulin requirement | 1 year
  Average daily insulin requirement
Beta cell function as assessed by beta-score | 1 year
  β-score is an assessment of beta cell function after islet transplantation incorporating fasting plasma glucose levels, HbA1c, daily insulin, and stimulated c-peptide. The range of the score is from 0 to 8. Higher number means better beta cell transplant function.

OTHER OUTCOMES:
Change in islet function between baseline to day 90±28 | 90 days
  Change in islet function between baseline to day 90±28. Islet function will be indicated by area under the curve of C-peptide levels during a mixed meal tolerance test adjusted by islet equivalent number transplanted.
Daily oral Morphine Equivalents on day prior to visit | 9 months
  Daily oral Morphine Equivalents on day prior to visit (day 90±28 to day 365±28)
Proportion of patients remaining on narcotics | 9 months
  Proportion of patients remaining on narcotics (day 90±28 to day 365±28).
Short form (SF)-12 Quality of Life score | 1 year
  SF-12 Quality of Life score, Scores range from 0 to100, with higher scores indicating better physical and mental healthy functioning.
Glycemic control measured by area under the curve (AUC) HbA1c through year 1 and the C-peptide AUC and HbA1c AUC through year 1 (measured every three months) as impacted in a multivariate model by the IEQ/kg islets transplanted. | 1 year
  Glycemic control measured by area under the curve (AUC) HbA1c through year 1 and the C-peptide AUC and HbA1c AUC through year 1 (measured every three months) as impacted in a multivariate model by the IEQ/kg islets transplanted.
Incidence and severity of adverse events and serious adverse events | 1 year
  Incidence and severity of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Charlton Strange, M.D, Study Director — Medical University of South Carolina; William Lancaster, M.D, Study Director — Medical University of South Carolina; Hongjun Wang, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Sutherland DE, Gruessner AC, Carlson AM, Blondet JJ, Balamurugan AN, Reigstad KF, Beilman GJ, Bellin MD, Hering BJ. Islet autotransplant outcomes after total pancreatectomy: a contrast to islet allograft outcomes. Transplantation. 2008 Dec 27;86(12):1799-802. doi: 10.1097/TP.0b013e31819143ec. PMID 19104425
- [Background] Morgan KA, Lancaster WP, Owczarski SM, Wang H, Borckardt J, Adams DB. Patient Selection for Total Pancreatectomy with Islet Autotransplantation in the Surgical Management of Chronic Pancreatitis. J Am Coll Surg. 2018 Apr;226(4):446-451. doi: 10.1016/j.jamcollsurg.2017.12.018. Epub 2017 Dec 28. PMID 29289751
- [Background] Wang J, Zhang Y, Cloud C, Duke T, Owczarski S, Mehrotra S, Adams DB, Morgan K, Gilkeson G, Wang H. Mesenchymal Stem Cells from Chronic Pancreatitis Patients Show Comparable Potency Compared to Cells from Healthy Donors. Stem Cells Transl Med. 2019 May;8(5):418-429. doi: 10.1002/sctm.18-0093. Epub 2019 Jan 24. PMID 30680957
- [Background] Song L, Sun Z, Kim DS, Gou W, Strange C, Dong H, Cui W, Gilkeson G, Morgan KA, Adams DB, Wang H. Adipose stem cells from chronic pancreatitis patients improve mouse and human islet survival and function. Stem Cell Res Ther. 2017 Aug 30;8(1):192. doi: 10.1186/s13287-017-0627-x. PMID 28854965
- [Background] Ryan EA, Paty BW, Senior PA, Lakey JR, Bigam D, Shapiro AM. Beta-score: an assessment of beta-cell function after islet transplantation. Diabetes Care. 2005 Feb;28(2):343-7. doi: 10.2337/diacare.28.2.343. PMID 15677790
- [Background] Wang H, Desai KD, Dong H, Owzarski S, Romagnuolo J, Morgan KA, Adams DB. Prior surgery determines islet yield and insulin requirement in patients with chronic pancreatitis. Transplantation. 2013 Apr 27;95(8):1051-7. doi: 10.1097/TP.0b013e3182845fbb. PMID 23411743